CLINICAL TRIAL: NCT03824548
Title: Real-World Analysis on the Diagnosis, Treatment Pattern and Outcomes for Patients With Gastro-Esophageal Reflux Disease (GERD) in China
Brief Title: Outcomes for Patients With Gastro-Esophageal Reflux Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Happy Life Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HLT-RWE-GERD-001
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Gastro-esophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: this is non-intervention study, there is no intervention drug or device in this study. — this is exactly a non-interventional study, no intervention during the whole study.

SUMMARY:
Gastro-esophageal reflux disease (GERD), the most common cause of erosive esophagitis (EE), remains highly prevalent worldwide.

GERD poses substantial burden on both patients and society. EE treatment patterns and unmet needs have been well-studied overseas, but evidence gaps still exist in China.

To fill these evidence gaps, real-world evidence for GERD and EE are needed. To understand GERD market we will analysis :Patient profile,GERD patient journey within hospital (first present, get diagnosed, receive initial and maintenance treatment),medication cost,department differentiation.

To investigate current treatment patterns of GERD / EE in China we will analysis: Current agents used and treatment duration in clinical practice treatment patterns by different reimbursement status treatment pattern by EE/NERD.

To get healing rate of EE we will analysis: Real-world efficacy of the current standard treatment (i.e. PPIs) for patient with two test results of gastroscopy.

The data required for this project are accessible in hospital electronic system; no specific data collection tools or methods are required for this project design. Only algorithms for retrieving and extracting eligible patients' records are required and will be developed by HLT based on the eligibility criteria defined in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Medical records of GERD, NERD and/or EE diagnoses （ICD code scope will be confirmed later）from January 1st, 2015 to December 31st, 2017.

oGERD is typically characterized by symptoms of heartburn and acid regurgitation. A diagnosis of EE or NERD can only be confirmed upon endoscopic examination.

* All ages, males or females
* A primary diagnosis of GERD/NERD/EE

For treatment patterns, patients are also required to have received one episode of treatment during the analysis period.

For RW treatment efficacy, the population will be restricted to the EE treatment population who underwent at least two endoscopy examinations.

Exclusion Criteria:

- No exclusion criteria will be applied for investigating diagnosis since all patients diagnosed with GERD, NERD, or EE should be captured regardless of whether they have medical conditions that affect their treatments.

A patient will not be eligible for investigating treatment patterns and RW treatment efficacy if he/she has any of the following exclusion criterion:

* A post-operative diagnosis of gastrointestinal cancers
* A diagnosis of esophageal foreign bodies or neoplasms
* A history of gastric or esophageal surgery
* Zollinger-Ellison syndrome
* Primary esophageal motility disorders (ex: achalasia)
* Esophageal strictures
* Eosinophilic esophagitis
* Identified as pregnant or lactating
* Hospitalized (inpatient) patients (to be confirmed by expert.) due to GERD as primary or secondary diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The overall analysis population will consist of patients of all ages who were diagnosed with GERD from January 2015 to December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of GERD patients with an EE diagnosis confirmed by physician judgment vs. endoscopy | oOnly patients diagnosed between January 1st, 2015 and October 31st, 2017 will be included to allow for at least an 8-week observational period.
  oAnalysis can be stratified by age group, sex, and health plan type to investigate possible differences in diagnostic practices based on these related patient characteristics.

SECONDARY OUTCOMES:
Similarly, descriptive statistics will also be presented for secondary endpoints as the analysis further examines treatment use and proxy indicators assessing real-world treatment efficacy. | Only patients diagnosed between January 1st, 2015 and October 31st, 2017 will be included to allow for at least an 8-week observational period.
  Proportion of EE patients and NERD patients by treatment use

CONTACTS AND LOCATIONS:
Locations (1):
- Yuan Na, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No